CLINICAL TRIAL: NCT00949624
Title: Phase I Study To Determine The Maximally Tolerated Dose Of Oral, Daily CP-868,596 And CP-868,596 Plus AG-013736 When Given In Combination With Docetaxel Administered Every 3 Weeks To Patients With Advanced Solid Tumors
Brief Title: CP-868,596 And CP-868,596 Plus AG-013736 In Combination With Docetaxel In Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arog Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5301005
Record Dates: First submitted 2009-07-24; First posted 2009-07-30 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2011-08

CONDITIONS: Advanced Solid Tumors
Keywords: PDGFr Inhibition;; VEGFr inhibition;; targeted therapy
MeSH Terms: interventions — crenolanib; Docetaxel; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): 60 mg BID/ 75 mg/m2
  Interventions: Drug: CP-868,596; Drug: Docetaxel
- Cohort 2 (Experimental): 100 mg BID/75 mg/m2
  Interventions: Drug: CP-868,596; Drug: Docetaxel
- Cohort 3 (Experimental): 100 mg BID/100 mg/m2
  Interventions: Drug: CP-868,596; Drug: Docetaxel
- Cohort 4b (Experimental): CP-868,596 + AG-013736 + TXT 75
  Interventions: Drug: CP-868,596; Drug: AG-013736; Drug: Docetaxel

INTERVENTIONS:
Drug: CP-868,596 — Oral tablet 60 mg BID continuous
  Arms: Cohort 1
Drug: Docetaxel — Intravenous 75 mg/m2 every three weeks
  Arms: Cohort 1
Drug: CP-868,596 — Oral tablet 100 mg BID continuous
  Arms: Cohort 2
Drug: Docetaxel — Intravenous 75 mg/m2 every three weeks
  Arms: Cohort 2
Drug: CP-868,596 — Oral tablet 100 mg BID continuous
  Arms: Cohort 3
Drug: Docetaxel — Intravenous 100 mg/m2 every three weeks
  Arms: Cohort 3
Drug: CP-868,596 — Oral tablet 60 mg BID continuous
  Arms: Cohort 4b
Drug: AG-013736 — Oral tablet 5 mg BID continuous
  Arms: Cohort 4b
Drug: Docetaxel — Intravenous 75 mg/m2 every three weeks
  Arms: Cohort 4b

SUMMARY:
A5301005 is a phase 1 study in patients with solid tumors which is testing the safety and tolerability of adding targeted agents to a standard chemotherapy. CP-868,596 is a platelet-derived growth factor receptor inhibitor (PDGFR) and AG-13736 is a vascular endothelial growth factor receptor inhibitor (VEGFR). This study will test the use of docetaxel (the standard chemotherapy) with either CP-868,596 or the combination of CP-868,596 and AG-13736.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥18 years old and with histologically or cytologically confirmed advanced solid tumors refractory/resistant to currently available therapies or for which there is no standard therapy.
* Patients with primary brain tumors are not eligible.
* Have at least one site of measurable disease.

Exclusion Criteria:

* Received chemotherapy (including targeted agents such as erlotinib), radiotherapy, immunotherapy or any investigational therapy within 3 weeks of study entry (within 6 weeks for previous treatments with nitrosoureas or mitomycin C).
* Received tamoxifen within 4 weeks prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
First-cycle Dose Limiting Toxicities | 2.5 years

SECONDARY OUTCOMES:
Determine the safety and tolerability of the combination of daily CP-868,596 and docetaxel on an every 3-week schedule | 2.5 years
Determine the safety and tolerability of the combination of daily CP-868,596 plus daily AG-013736 plus docetaxel on an every 3-week schedule | 2.5 years
To evaluate the pharmacokinetics (PK) of CP-868,596 and docetaxel when given in combination | 2.5 years
To evaluate the pharmacokinetics (PK) of CP-868,596, AG-013736 and docetaxel when given in combination | 2.5 years
Conduct biomarker investigations on plasma/serum samples to explore critical events in pharmacodynamic response to CP-868,596 (eg, VEGF, phospho-SHP, etc.) | 2.5 years
To explore the relationship between polymorphisms in genes involved in the metabolism and transport of CP-868,596 and pharmacokinetic/pharmacodynamic parameters | 2.5 years
To explore the effects of CP-868,596 on tumor blood flow and permeability via DCE-MRI | 2.5 years
To assess any preliminary clinical evidence of anti-tumor activity using RECIST | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Pfizer Investigational Site, Durham, North Carolina, United States
- Pfizer Investigational Site, East Melbourne, Victoria, Australia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5301005&StudyName=CP-868%2C596%20And%20CP-868%2C596%20Plus%20AG-013736%20In%0ACombination%20With%20Docetaxel%20In%20Advanced%20Solid%20Tumors%0A